CLINICAL TRIAL: NCT01513954
Title: Examination of Serum Progesterone Levels in an IVF Population Following Two Types of Egg Aspiration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Red Rock Fertility Center (Other)
Collaborators: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 20111821
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Infertility, Female
Keywords: Infertility
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IVF population: Long Lupron IVF Population
- IUI patients: Patients undergoing IUI

SUMMARY:
The purpose of this study is to determine whether progesterone hormone levels differ following egg retrieval with a single lumen needle compared with a double lumen needle. These levels will be measured on several days before and after egg retrieval. The progesterone levels in each IVF group will also be compared to the group of women who are having IUI. In addition, these progesterone levels will be correlated with pregnancy outcomes.

DETAILED DESCRIPTION:
This is a prospective randomized trial consisting of 3 groups of patients. Following a long lupron protocol IVF cycle there is a need for supplemental progesterone. The purpose of this study is to determine what range of serum levels should be observed when differing methods of egg aspiration have been administered and whether or not there is a correlation with outcomes or pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 21-37
* Cycle Day 3 FSH between 2-12
* History of regular menstrual cycles between 24-34 days

Exclusion Criteria:

* Previous IVF failure
* Severe male factor
* Severe obesity, BMI > 40
* More than 20 follicles on ultrasound prior to retrieval

Ages: 21 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: IUI patients and IVF patients following a long lupron protocol cycle
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eva D Littman, M.D., Principal Investigator — Red Rock Fertility Center
Locations (1):
- Red Rock Fertility Center, Las Vegas, Nevada, United States